CLINICAL TRIAL: NCT04439929
Title: A Randomized, Double-blind, Two-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Two Formulations of Adalimumab (TUR01 and EU Sourced Humira®) in Healthy Subjects
Brief Title: Comparative Pharmacokinetic, Safety, Tolerability and Immunogenicity Study of Adalimumab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turgut İlaçları A.Ş. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 240648
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Healthy Participants
Keywords: adalimumab; biosimilar; healthy; phase 1; pharmacokinetics; bioequivalence
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab-TUR01 (Experimental)
  Interventions: Biological: TUR01
- Adalimumab-EU (Active Comparator)
  Interventions: Biological: Adalimumab-EU

INTERVENTIONS:
Biological: TUR01 — Administered as a single 40 mg, subcutaneous dose
  Other Names: Adalimumab-Turgut
  Arms: Adalimumab-TUR01
Biological: Adalimumab-EU — Administered as a single 40 mg, subcutaneous dose
  Other Names: Humira
  Arms: Adalimumab-EU

SUMMARY:
This is a randomized, double-blind, two-arm, parallel group, single-dose study to demonstrate pharmacokinetic, safety, tolerability and immunogenicity similarity of biosimilar candidate TUR01 to EU-sourced Humira® in healthy participants after administration of adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential or healthy male subjects aged 18 to 55 years (inclusive at screening).
* Have body weight between 65.0 to 90.0 kg and a body mass index between 20.0 to 29.9 kg/m2, inclusive.
* Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
* Must be able to provide written informed consent, which must be obtained prior to any study related procedures.

Exclusion Criteria:

* Evidence or history of clinically significant or relevant pathology.
* Have either active or latent tuberculosis.
* Have received treatment with a monoclonal antibody or fusion protein within 9 months prior to administration and/or have evidence of immunogenicity from previous exposure to a monoclonal antibody or fusion protein.
* Have a mental disease classified as serious by the Investigator.
* Have received live vaccine(s) within 4 weeks prior to Screening or who will require live vaccine(s) between Screening and the final study visit.
* Who intake alcoholic beverages more than 28 units per week.
* Have taken medication with a half-life of > 24 h within 4 weeks or 10 half-lives of the medication prior to investigational medicinal product administration.
* Have donated > 100 mL of blood or plasma within 4 weeks prior to investigational medicinal product administration.
* Have participated in another study with an investigational drug within 4 weeks prior to investigational medicinal product administration. Subjects who have received treatment with a biological or immunosuppressive agent within 3 months of screening should also be excluded.
* Subjects who are not able to consume standardized meals provided by the clinical study site during hospitalization.
* Subjects who, in the opinion of the Investigator, are not likely to complete the study for whatever reason.
* Involvement of any sponsor, study site/contract research organisation employee, Investigator or their close relatives.
* Vulnerable subjects.
* Pregnant or nursing women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUCinf) | Day 1 - Day 71
  AUCinf = area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) + last observed concentration (Ct)/terminal rate constant (λz)
Maximum serum concentration (Cmax) | Day 1 - Day 71
  Cmax

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) | Day 1 - Day 71
Area under the concentration-time curve from time zero to 336 hours (AUC336) | Day 1 - Day 15
  Area under the concentration-time curve from time zero to 14 days
Area under the concentration-time curve from time zero to 672 hours (AUC672) | Day 1 - Day 29
  Area under the concentration-time curve from time zero to 28 days
Area under the concentration-time curve from time zero to 1008 hours (AUC1008) | Day 1 - Day 43
  Area under the concentration-time curve from time zero to 42 days
Area under the concentration-time curve from time zero to 1680 hours (AUC1680) | Day 1 - Day 71
  Area under the concentration-time curve from time zero to 70 days
Time to Cmax (Tmax) | Day 1 - Day 71
  Time to reach the maximum concentration
Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 - Day 71
Terminal rate constant (λz) | Day 1 - Day 71
  The parameter will be calculated by linear least squares regression analysis using at least 3 non-zero concentrations in the terminal phase
Terminal half-life calculated by ln(2)/λz (t½) | Day 1 - Day 71
Apparent total body clearance (CL/F) | Day 1 - Day 71
Area under the concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCextrap) | Day 1 - Day 71

OTHER OUTCOMES:
Immunogenicity - Incidence of anti-drug antibodies to adalimumab | Day 1 - Day 71
Immunogenicity - Incidence of neutralizing antibodies | Day 1 - Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- PAREXEL International GmbH, Early Phase Clinical Unit Berlin, Berlin, Germany